CLINICAL TRIAL: NCT03415672
Title: Immunogenicity and Safety of HBAI20 Hepatitis B Vaccine in Non-responders
Brief Title: Hepatitis B Vaccine for Non-responders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: CyTuVax (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HBnr02; 2016-002720-91 (EudraCT Number)
Record Dates: First submitted 2018-01-05; First posted 2018-01-30 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Hepatitis B
Keywords: Interleukin-2; Hepatitis B Vaccines; Non-responders; Liver Diseases; Digestive system; Vaccines
MeSH Terms: conditions — Hepatitis B; Liver Diseases | interventions — Hepatitis B Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Subjects included in Group 1 are adults who are non-responders (did not achieve seroprotection after 3 or more vaccinations with a Hepatitis B vaccine. They will receive three doses of HBVaxPro-10μg at 0, 1, and 2 months. The HBVaxPro-10μg vaccines are administered strictly intramuscularly in the deltoid muscle and must not be injected intravascularly.
  Interventions: Biological: HBVaxPro
- Group 2 (Experimental): Subjects included in Group 2 are adults who are non-responders (did not achieve seroprotection after 3 or more vaccinations with a Hepatitis B vaccine). They will receive three doses of HBAI20 at 0, 1, and 2 months.
  The HBAI20 vaccines are administered strictly intramuscularly in the deltoid muscle and must not be injected intravascularly.
  Interventions: Biological: HBAI20

INTERVENTIONS:
Biological: HBVaxPro — Three doses of HBVaxPro-10μg at 0, 1, and 2 months. The HBVaxPro-10μg vaccines are administered strictly intramuscularly in the deltoid muscle and must not be injected intravascularly.
  Arms: Group 1
Biological: HBAI20 — Three doses of HBAI20 at 0, 1, and 2 months. The HBAI20 vaccines are administered strictly intramuscularly in the deltoid muscle and must not be injected intravascularly.
  Arms: Group 2

SUMMARY:
In the current study, the investigators study the efficacy of the HBAI20 vaccine to induce seroprotection in registered non-responders (adults who were previously vaccinated with the HBVaxPro-10μg but did not achieve seroprotection). The study will further assess the safety of the HBAI20 vaccine in comparison with HBVaxPro-10μg.

DETAILED DESCRIPTION:
Rationale:

Worldwide, people are suffering from the consequences of Hepatitis B (HB) virus infection. Currently available vaccines are protective in most of the vaccinees, however, a small part of the population does not respond to these vaccines (non-responders). A new adjuvant (AI20) has been developed by CyTuVax to improve the standard Hepatitis B vaccine for the protection of non-responders. The AI20 adjuvant consists of depot-attached rhuIL-2 (aggregated Interleukin-2 (IL-2) molecules attached to alum), facilitating the slow release of highly concentrated IL-2 nano aggregates. In preclinical experiments, vaccination of mice, rats, and rabbits with the new HBAI20 vaccine results in higher and earlier immune responses to HBsAg compared to vaccination with one of the standard Hepatitis B vaccines. The phase 1 clinical trial showed that the HBAI20 vaccine was well tolerated and it induced protective anti Hepatitis B antibody titers in 9 out of 10 non-responders (subjects vaccinated at least 6 times with the Hepatitis B vaccine). The phase 2 clinical trial will be conducted in order to assess the immunogenicity and safety of the AI20 adjuvant and further test if the AI20 adjuvanted Hepatitis B vaccine induces protective antibody titers in the vaccinated non-responders.

Objective: In the current study, the investigators study the efficacy of the HBAI20 vaccine to induce seroprotection. Furthermore, the investigators will compare the safety of the HBAI20 vaccine with the HBVaxPro-10μg.

Study design:

Multicenter double blinded randomized controlled intervention phase II study.

Study population:

Registered non-responders after at least 3 HBV vaccinations (n=132- 140) 18-59 years of age, males and females.

Intervention:

The study will include 2 groups. HB vaccine registered non-responder subjects after at least 3 vaccinations are randomized into group 1 (n= 33 to 35) or 2 (n= 99 to 105) at a 1 to 3 ratio. No less than 40% of the subjects of each group should have received only 1 series of Hepatitis B vaccination. "Group 1" subjects receive the standard HB vaccine (HBVaxPro-10μg) and "Group 2" subjects receive the HBAI20 vaccine. All study subjects will receive 3 vaccinations separated by one month (0, 1, and 2 months) in accordance with the recommended vaccination schedule for non-responders in the Netherlands.

Main study parameters/endpoints:

The primary study parameter is the immunogenicity of the adjuvanted vaccine. The immunogenicity of the adjuvanted vaccine is measured as the percentage of subjects that attain seroprotection after the first vaccination at 1, 2, and 3,5 months (HBsAg antibodies ≥10 mIU/ml measure by the COBAS system). The secondary study parameter is the safety of the vaccination. The safety of the vaccination is the number and severity of the local and systemic adverse reactions.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Study subjects will be vaccinated 3 times at 0, 1, and 2 months from the beginning of the study and invited to the hospital or vaccination centre for 4 or 5 visits. The risks associated with participation in this study are considered to be low and comparable with standard vaccines. Physical discomfort after vaccine administration can occur at the injection site (redness, swelling, etc.) and systemically (fever, fatigue, headache). Effects are expected to occur for a short period of time (within the first 4 days after the first and second injection). In addition subjects may experience adverse reactions to the cytokine component of the adjuvant. Because of the very low dose of the cytokine component of the adjuvant, which will be gradually released, the risks are expected to be low. The potential risks of venepuncture for blood sampling are mild pain and haematoma, and are considered low. Subjects may benefit from this study by becoming immunized (seroprotected) against Hepatitis B. Becoming seroprotected is important for the non-responder subjects because most of the registered non-responders are healthcare workers who can be exposed to the Hepatitis B virus.

ELIGIBILITY:
Inclusion Criteria:

* In good health as determined by the outcome of medical history, physical examination screening/baseline labs and clinical judgment of the clinical investigator
* Age 18 to 59 years, inclusive at the time of enrollment
* Willing and able to adhere to the study regimen
* Willing to adhere to a highly effective birth control method during the duration of the study
* Having a signed informed consent form
* Documented non-responders: Subjects with documented one or more cycles of Hepatitis B vaccination (total of 3 or more vaccinations) and titer analysis 1 to 3 months after the last vaccination that show that they have not developed the Hepatitis B antibody titer recommended after standard vaccination: HBsAg antibody titer superior to 10mIU/ml. In case the subjects do not have a titer analysis performed 1 to 3 months after their last recorded vaccination, the potential subject can be included after permission from the project leader after analysis of the case file.

Exclusion Criteria:

* Any infectious disease at the time of screening and/or enrollment
* Positive HIV, Hepatitis B virus or Hepatitis C virus serology
* Known or suspected immune deficiency
* Known or suspected disease that influences the immune system including chronic allergies that require frequent anti-allergy medication - excluding anti-histaminics -, cancer and transplantation recipients
* Known or suspected allergy to any of the vaccine components
* Dialysis patient
* History of unusual or severe reactions to any previous vaccination
* History of any neurologic disorder, including epilepsy and autism
* Use of medication that influences the immune system (immune suppressive treatment or daily use of corticosteroids, including chronic use of local corticosteroids)
* Any vaccination within 3 months before screening excluding flu vaccination
* Blood donation within 1 month before screening
* Administration of plasma (incl. immunoglobulins) or blood products within 12 months before screening
* Participation in another clinical trial within 3 months before screening
* Abnormal pre-treatment laboratory parameters which are clinically relevant according to the investigator
* Bleeding disorders. Participants on coumadins anticoagulants and participants receiving 2 platelet aggregation inhibitors can not be included in the study. People on the direct oral anticoagulant dabigatran, apixaban, edoxaban, and rivaroxaban and participants using only one platelet aggregation inhibitor can be included.
* Female subjects planning to become pregnant or breastfeeding babies until visit 4
* Females: positive pregnancy test at screening date
* Excessive alcohol or controlled drug use - More than 2 alcohol measures per day (one alcohol measure is a beer (250ml) or one glass of wine (125ml) or one strong measure (35ml) or one port/sherry (75ml)). Regular use of controlled drugs
* Any Hepatitis B vaccination in the last 3 months Temporary exclusion criterion for vaccination
* Temperature > 38.4°C will lead to postponement of participation and vaccination.

Screening may continue when the temperature has normalized.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 133 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2019-01-09 (Actual); Study Completion 2019-01-09 (Actual)

PRIMARY OUTCOMES:
Immunogenicity of the HBAI20 | Six weeks after the third vaccination.
  Anti Hepatitis B surface antigen antibody titer.

SECONDARY OUTCOMES:
Safety of the HBAI20 Hepatitis B vaccine: Percentage of subjects reporting adverse events after being vaccinated. | The whole duration of the study protocol (102 days)
  Percentage of subjects reporting adverse events after being vaccinated.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre van Damme, MD, PhD, Principal Investigator — Vaxinfectio - Antwerp University; Geert Robaeys, MD, PhD, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (3):
- Belgium (2):
  - Vaxinfectio - Antwerp University, Antwerp
  - Ziekenhuis Oost-Limburg, Genk
- Maastricht UMC, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Coates T, Wilson R, Patrick G, Andre F, Watson V. Hepatitis B vaccines: assessment of the seroprotective efficacy of two recombinant DNA vaccines. Clin Ther. 2001 Mar;23(3):392-403. doi: 10.1016/s0149-2918(01)80044-8. PMID 11318074
- [Background] Jack AD, Hall AJ, Maine N, Mendy M, Whittle HC. What level of hepatitis B antibody is protective? J Infect Dis. 1999 Feb;179(2):489-92. doi: 10.1086/314578. PMID 9878036
- [Background] Yu AS, Cheung RC, Keeffe EB. Hepatitis B vaccines. Infect Dis Clin North Am. 2006 Mar;20(1):27-45. doi: 10.1016/j.idc.2006.01.004. PMID 16527647
- [Background] Cardell K, Akerlind B, Sallberg M, Fryden A. Excellent response rate to a double dose of the combined hepatitis A and B vaccine in previous nonresponders to hepatitis B vaccine. J Infect Dis. 2008 Aug 1;198(3):299-304. doi: 10.1086/589722. PMID 18544037
- [Background] Halperin SA, Dobson S, McNeil S, Langley JM, Smith B, McCall-Sani R, Levitt D, Nest GV, Gennevois D, Eiden JJ. Comparison of the safety and immunogenicity of hepatitis B virus surface antigen co-administered with an immunostimulatory phosphorothioate oligonucleotide and a licensed hepatitis B vaccine in healthy young adults. Vaccine. 2006 Jan 9;24(1):20-6. doi: 10.1016/j.vaccine.2005.08.095. Epub 2005 Sep 12. PMID 16198027
- [Background] Halperin SA, Ward BJ, Dionne M, Langley JM, McNeil SA, Smith B, Mackinnon-Cameron D, Heyward WL, Martin JT. Immunogenicity of an investigational hepatitis B vaccine (hepatitis B surface antigen co-administered with an immunostimulatory phosphorothioate oligodeoxyribonucleotide) in nonresponders to licensed hepatitis B vaccine. Hum Vaccin Immunother. 2013 Jul;9(7):1438-44. doi: 10.4161/hv.24256. Epub 2013 Apr 9. PMID 23571179
- [Background] Ambrosch F, Wiedermann G, Kundi M, Leroux-Roels G, Desombere I, Garcon N, Thiriart C, Slaoui M, Thoelen S. A hepatitis B vaccine formulated with a novel adjuvant system. Vaccine. 2000 Apr 14;18(20):2095-101. doi: 10.1016/s0264-410x(99)00566-6. PMID 10715523
- [Background] Levie K, Gjorup I, Skinhoj P, Stoffel M. A 2-dose regimen of a recombinant hepatitis B vaccine with the immune stimulant AS04 compared with the standard 3-dose regimen of Engerix-B in healthy young adults. Scand J Infect Dis. 2002;34(8):610-4. doi: 10.1080/00365540110080881. PMID 12238579
- [Background] Desombere I, Van der Wielen M, Van Damme P, Stoffel M, De Clercq N, Goilav C, Leroux-Roels G. Immune response of HLA DQ2 positive subjects, vaccinated with HBsAg/AS04, a hepatitis B vaccine with a novel adjuvant. Vaccine. 2002 Jun 7;20(19-20):2597-602. doi: 10.1016/s0264-410x(02)00150-0. PMID 12057618
- [Background] Jacques P, Moens G, Desombere I, Dewijngaert J, Leroux-Roels G, Wettendorff M, Thoelen S. The immunogenicity and reactogenicity profile of a candidate hepatitis B vaccine in an adult vaccine non-responder population. Vaccine. 2002 Nov 1;20(31-32):3644-9. doi: 10.1016/s0264-410x(02)00397-3. PMID 12399191
- [Background] Pocock SJ, Simon R. Sequential treatment assignment with balancing for prognostic factors in the controlled clinical trial. Biometrics. 1975 Mar;31(1):103-15. PMID 1100130
- [Background] Siegel JP, Puri RK. Interleukin-2 toxicity. J Clin Oncol. 1991 Apr;9(4):694-704. doi: 10.1200/JCO.1991.9.4.694. PMID 2066765
- [Background] Vial T, Descotes J. Clinical toxicity of interleukin-2. Drug Saf. 1992 Nov-Dec;7(6):417-33. doi: 10.2165/00002018-199207060-00004. PMID 1418698